CLINICAL TRIAL: NCT07358494
Title: Effect of Diluted Thyme Honey On Dry Mouth In Intensive Care Unit Patients Exposed to Oxygen Flow Therapy: A Randomized Controlled Study
Brief Title: Effect of Diluted Thyme Honey On Dry Mouth In Intensive Care Unit Patients Exposed to Oxygen Flow Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esra Yaprak Gokturk (Other)
Responsible Party: Sponsor-Investigator, Esra Yaprak Gokturk, MSN: Master of Science in Nursing, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AnkaraU-esrayaprakgokturk01
Record Dates: First submitted 2025-05-21; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Nursing Care
Keywords: Xerostomia; Thyme Honey; Nursing; Nasal Oxygen Flow Treatment
MeSH Terms: conditions — Xerostomia | interventions — Mouthwashes

STUDY DESIGN:
Intervention Model Description: This study has a randomized controlled experimental design.
Who Masked: Participant, Care Provider
Masking Description: Randomization Participants included in the study were assigned to the intervention or control groups using a simple randomization method involving envelopes. Numbers ranging from 1 to 64, representing patient numbers, were automatically distributed at random via the website https://www.calculatorsoup.com/calculators/statistics/random-number-generator.php, thereby creating "Set 1." It was determined that the first 32 of the 64 randomly arranged numbers in 'Set 1' would represent patients in the intervention group, and the last 32 would represent patients in the control group.
  After obtaining consent from the patients participating in the study, they were asked to draw one sealed envelope from a bag containing sealed envelopes with numbers from 1 to 64 written on them. The envelopes drawn by the patients were opened in their presence. The researcher determined which group the patients would be included in, either the intervention or control group, based on the number that came out of the
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diluted thyme honey arm (Experimental): * After obtaining informed consent from participants who agreed to participate in the study, they were asked to draw one sealed envelope from a bag containing sealed envelopes numbered from 1 to 64. The envelopes drawn by the patients were opened in their presence. The researcher determined whether the patients would be included in the intervention or control group based on the number drawn from the envelope.
  * Participants assigned to the intervention group were first given the Patient Information Form. Then, before starting the intervention, participants were asked questions from the "Subjective Dry Mouth Assessment Form" prepared by Duruk (2012) using the Visual Analogue Scale. Each point given in response to the questions was recorded in the Patient Follow-up Form.
  * Patients were educated on the importance of dry mouth, the types of foods and liquids to avoid, the necessity of adequate saliva secretion, the functions of saliva, methods of coping with dry mouth, and the necess
  Interventions: Other: diluted thyme honey arm; Other: Mouth wash
- 0.9% NaCl arm (Placebo Comparator): After obtaining informed consent from participants who agreed to participate in the study, they were asked to draw one sealed envelope from a bag containing sealed envelopes with numbers ranging from 1 to 64 written on them. The envelopes drawn by the patients were opened in their presence. Patients were assigned to either the intervention or control group according to the number drawn from the envelope.
  * Participants in the control group were first given the Patient Information Form. Then, before starting the application, they were asked questions from the Subjective Dry Mouth Assessment Form. Each point given in response to the questions was recorded in the Patient Follow-up Form.
  * Patients were educated on the importance of dry mouth, the types of foods and liquids to avoid, the necessity of adequate saliva secretion, the functions of saliva, methods for coping with dry mouth, and the necessary precautions to identify and report any side effects that
  Interventions: Other: Mouth wash

INTERVENTIONS:
Other: diluted thyme honey arm — In this study, the feasibility of an alternative method for alleviating dry mouth, which is very important in terms of nursing care, was investigated. The effect of diluted thyme honey, which had not been previously studied, on dry mouth was investigated in intensive care patients receiving nasal oxygen flow therapy in the intervention group. The control group received oral care using a standard oral care solution of 0.9% NaCl.
  Arms: diluted thyme honey arm
Other: Mouth wash — In this study, the usability of an alternative method for the elimination of dry mouth, which has a very important place in terms of nursing care, was investigated. The effect of diluted thyme honey on dry mouth in intensive care patients receiving nasal oxygen flow therapy, which has not been previously studied in the literature, was investigated.

SUMMARY:
This research is a randomized, controlled, double-blind, experimental study conducted to investigate the effect of diluted thyme honey on dry mouth in individuals receiving treatment in intensive care and receiving nasal oxygen flow therapy.

H0: There is no significant difference in reducing dry mouth in intensive care patients receiving nasal oxygen flow therapy between the intervention group receiving oral care with diluted thyme honey and the control group receiving standard oral care.

The study sample consisted of 64 inpatients receiving nasal oxygen flow therapy in the Emergency Intensive Care and Emergency Critical Intensive Care Units of Ankara Training and Research Hospital. Patients were divided into groups using a sealed envelope method. Patients in the intervention group received oral care using diluted thyme honey, while patients in the control group received oral care using 0.9% NaCl.

DETAILED DESCRIPTION:
SUMMARY

Backround Dry mouth due to nasal oxygen flow therapy is one of the side effects frequently experienced by patients treated in intensive care units. Although there are various pharmacological and complementary medicine methods for the prevention and treatment of dry mouth, this condition continues to negatively affect the daily lives of patients due to the lack of a definitive method and the neglect of oral care.

Aim The aim of this study was to evaluate the efficacy of diluted thyme honey in preventing dry mouth in intensive care patients receiving nasal oxygen flow therapy.

Desing This study has a randomized controlled experimental design.

Methods This study included 64 intensive care unit patients receiving nasal oxygen flow therapy. It was a randomized controlled experimental study consisting of intervention (thyme honey) and control group (0.9% NaCl). Participants were randomized to the groups by closed envelope method. 32 patients were included in both groups. Patients in both groups included in the study underwent the same protocol steps except for the oral care product (thyme honey and 0.9% NaCl). After obtaining consent from the patients who agreed to be included in the study, information about the participants was collected by asking the Patient Information Form prepared by the researcher. The Subjective Dry Mouth Form was administered to the participants before the start of the study and at the end of the 3rd day when the application protocols were completed. After the applications were completed, the pre-test and post-test scores of the patients in response to each question in the 'Subjective Dry Mouth Evaluation Form' and their answers to an open-ended question about their opinions on thyme honey in the Patient Information Form were combined in the patient follow-up form.

ELIGIBILITY:
Inclusion Criteria:

* Being treated under intensive care conditions and receiving nasal oxygen flow therapy above 4L/min,
* Over 18 years of age,
* Not diagnosed with Sjögren's Syndrome,
* No previous exposure to radiotherapy or chemotherapy,
* Has not had a salivary gland infection,
* Has not undergone an operation to remove the salivary glands,
* Not allergic to honey,
* No chewing or swallowing difficulties,
* Not using thyme-containing products for oral care in the previous period,
* Patients who did not have any communication problems and who voluntarily agreed to participate in the study were included in the study

Exclusion Criteria:

- Patients who did not meet the inclusion criteria and did not voluntarily agree to participate in the study were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The Effect of Diluted Thyme Honey on Dry Mouth in Intensive Care Patients Receiving Nasal Oxygen Flow Therapy: A Randomized Controlled Trial | 9 week
  The Subjective Dry Mouth Assessment Form was used to assess dry mouth. This form includes questions regarding symptoms such as "dry mouth," "difficulty swallowing," "difficulty speaking," "waking up from sleep," "dry tongue," "burning mouth," "burning throat," "dry throat," "thirst," "bad taste in the mouth," "saliva volume," and "bad breath." Responses are scored on a 0-10 scale using 11 Visual Analogue Scales (VAS). Scoring begins with 0 (not at all) and ends with 10 (extremely).
  The Subjective Dry Mouth Assessment Form was administered to patients before the study began to gather patient information and determine their dry mouth levels. At the end of the third day, the Subjective Dry Mouth Assessment Form was administered to the patients, who underwent three days of treatment, and their dry mouth was re-evaluated. Data on the patients' dry mouth levels were collected before and after the study.

CONTACTS AND LOCATIONS:
Overall Officials: ayten demir, assoc.prof.dr., Study Director — Ankara University
Locations (1):
- Ankara University Institute of Health Sciences Department of Nursing, Ankara, Dışkapı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] YAVUZ KARAMANOĞLU A, YAVUZ M (2015). Ağız Sağlığı Hemşirelik Değerlendirmesinde Kanıtlar Ve Uygulama Önerileri. Ege Üniversitesi Hemşirelik Fakültesi Dergisi, 31(1): 131-143.
- [Result] Takzaree N, Hassanzadeh G, Rouini MR, Manayi A, Hadjiakhondi A, Majidi Zolbin M. Evaluation of the Effects of Local Application of Thyme Honey in Open Cutaneous Wound Healing. Iran J Public Health. 2017 Apr;46(4):545-551. PMID 28540272
- [Result] TABACHNICK B G, FIDELL L S, (2013). Using multivariate statistics. Boston:Pearson. 6: 497-516.
- [Result] SEO E, SONG J, HUR M, LEE M, SOO LEE M (2017). Effects of aroma mouthwash on stress level, xerostomia, and halitosis in healthy nurses: A non-randomized controlled clinical trial. European Journal of Integrative Medicine, 10: 82-89. DOI: 10.1016/j.eujim.2017.03.001
- [Result] ÖZKÖK A, KORU Ö, SORKUN K (2016). Microbiological Analysis And Antibacterial Effects Of Turkish Thyme Honey. Bee World, 93(4): 98-101. DOI: 10.1080/0005772X.2016.1275489
- [Result] Lopez-Pintor RM, Casanas E, Gonzalez-Serrano J, Serrano J, Ramirez L, de Arriba L, Hernandez G. Xerostomia, Hyposalivation, and Salivary Flow in Diabetes Patients. J Diabetes Res. 2016;2016:4372852. doi: 10.1155/2016/4372852. Epub 2016 Jul 10. PMID 27478847
- [Result] Li Y, Taylor JM, Ten Haken RK, Eisbruch A. The impact of dose on parotid salivary recovery in head and neck cancer patients treated with radiation therapy. Int J Radiat Oncol Biol Phys. 2007 Mar 1;67(3):660-9. doi: 10.1016/j.ijrobp.2006.09.021. Epub 2006 Dec 4. PMID 17141973
- [Result] Lagerlof F, Dawes C. The volume of saliva in the mouth before and after swallowing. J Dent Res. 1984 May;63(5):618-21. doi: 10.1177/00220345840630050201. PMID 6584462
- [Result] Lafraxo H, Bakour M, Laaroussi H, El Ghouizi A, Ousaaid D, Aboulghazi A, Lyoussi B. The Synergistic Beneficial Effect of Thyme Honey and Olive Oil against Diabetes and Its Complications Induced by Alloxan in Wistar Rats. Evid Based Complement Alternat Med. 2021 Sep 20;2021:9949056. doi: 10.1155/2021/9949056. eCollection 2021. PMID 34594393
- [Result] Konings AW, Coppes RP, Vissink A. On the mechanism of salivary gland radiosensitivity. Int J Radiat Oncol Biol Phys. 2005 Jul 15;62(4):1187-94. doi: 10.1016/j.ijrobp.2004.12.051. PMID 15990024
- [Result] Kobya Bulut H, Guducu Tufekci F. Honey prevents oral mocositis in children undergoing chemotherapy: A quasi-experimental study with a control group. Complement Ther Med. 2016 Dec;29:132-140. doi: 10.1016/j.ctim.2016.09.018. Epub 2016 Sep 19. PMID 27912937
- [Result] KILAVUZ, DERVİŞ KAAN (2014). Türk Toplumunda Ağız Kuruluğu Prevalansının Araştırılması. Doktora Tezi, Gazi Üniversitesi.
- [Result] Kannarkat G, Lasher EE, Schiff D. Neurologic complications of chemotherapy agents. Curr Opin Neurol. 2007 Dec;20(6):719-25. doi: 10.1097/WCO.0b013e3282f1a06e. PMID 17992096
- [Result] Hashemian F, Baghbanian N, Majd Z, Rouini MR, Jahanshahi J, Hashemian F. The effect of thyme honey nasal spray on chronic rhinosinusitis: a double-blind randomized controlled clinical trial. Eur Arch Otorhinolaryngol. 2015 Jun;272(6):1429-35. doi: 10.1007/s00405-014-3233-x. Epub 2014 Aug 9. PMID 25106547
- [Result] Hanchanale S, Adkinson L, Daniel S, Fleming M, Oxberry SG. Systematic literature review: xerostomia in advanced cancer patients. Support Care Cancer. 2015 Mar;23(3):881-8. doi: 10.1007/s00520-014-2477-8. Epub 2014 Oct 18. PMID 25322971
- [Result] GEORGE D, MALLERY M (2010). SPSS for Windows Step by Step: A Simple Guide and Reference, 17.0 update (10a ed.) Boston: Pearson
- [Result] Ganjre A, Kathariya R, Bagul N, Pawar V. Anti-carcinogenic and Anti-bacterial Properties of Selected Spices: Implications in Oral Health. Clin Nutr Res. 2015 Oct;4(4):209-15. doi: 10.7762/cnr.2015.4.4.209. Epub 2015 Oct 31. PMID 26566515
- [Result] Fantozzi PJ, Pampena E, Di Vanna D, Pellegrino E, Corbi D, Mammucari S, Alessi F, Pampena R, Bertazzoni G, Minisola S, Mastroianni CM, Polimeni A, Romeo U, Villa A. Xerostomia, gustatory and olfactory dysfunctions in patients with COVID-19. Am J Otolaryngol. 2020 Nov-Dec;41(6):102721. doi: 10.1016/j.amjoto.2020.102721. Epub 2020 Sep 10. PMID 32977063
- [Result] DURUK NAZİKE (2012). Hemodiyaliz Sırasında Ciklet Çiğnemenin Ağız Kuruluğu Ve Semptomlarına Etkisi. Doktora Tezi, Ege Üniversitesi.
- [Result] DAVIES A N. EPSTEIN J B (2010). Salivary gland dysfunction Oral Complications of Cancer and its Management. Oxford University Press, p: 203-223. DOI: 10.1016/j.gerinurse.2015.10.014
- [Result] Dalodom S, Lam-Ubol A, Jeanmaneechotechai S, Takamfoo L, Intachai W, Duangchada K, Hongsachum B, Kanjanatiwat P, Vacharotayangul P, Trachootham D. Influence of oral moisturizing jelly as a saliva substitute for the relief of xerostomia in elderly patients with hypertension and diabetes mellitus. Geriatr Nurs. 2016 Mar-Apr;37(2):101-9. doi: 10.1016/j.gerinurse.2015.10.014. Epub 2015 Nov 26. PMID 26631691
- [Result] Crogan NL. Managing xerostomia in nursing homes: pilot testing of the Sorbet Increases Salivation intervention. J Am Med Dir Assoc. 2011 Mar;12(3):212-6. doi: 10.1016/j.jamda.2010.06.002. Epub 2010 Oct 8. PMID 21333924
- [Result] Chanques G, Constantin JM, Sauter M, Jung B, Sebbane M, Verzilli D, Lefrant JY, Jaber S. Discomfort associated with underhumidified high-flow oxygen therapy in critically ill patients. Intensive Care Med. 2009 Jun;35(6):996-1003. doi: 10.1007/s00134-009-1456-x. Epub 2009 Mar 18. PMID 19294365
- [Result] Charalambous M, Raftopoulos V, Paikousis L, Katodritis N, Lambrinou E, Vomvas D, Georgiou M, Charalambous A. The effect of the use of thyme honey in minimizing radiation - induced oral mucositis in head and neck cancer patients: A randomized controlled trial. Eur J Oncol Nurs. 2018 Jun;34:89-97. doi: 10.1016/j.ejon.2018.04.003. Epub 2018 Apr 30. PMID 29784145
- [Result] Charalambous A, Lambrinou E, Katodritis N, Vomvas D, Raftopoulos V, Georgiou M, Paikousis L, Charalambous M. The effectiveness of thyme honey for the management of treatment-induced xerostomia in head and neck cancer patients: A feasibility randomized control trial. Eur J Oncol Nurs. 2017 Apr;27:1-8. doi: 10.1016/j.ejon.2017.01.001. Epub 2017 Jan 16. PMID 28279391
- [Result] BORAHAN, M.OĞUZ (2005). Anksiyete, Depresyon, Stres ve Medikasyonun Tükürük Akış Hızı ve Subjektif Ağız Kuruluğu Üzerine Olan Etkilerinin İncelenmesi. Doktora Tezi, Marmara Üniversitesi.
- [Result] BİLGE M, TOZOĞLU Ü, 2022. Diyabetes Mellitus Olgularında Oral Mukoza Bulguları. Duzce Medical Journal, 12(2): 12 - 16.
- [Result] BİÇİCİ, BERNA (2010). Mcgill Ağrı Ölçeği Kısa Formu"nun Geçerlik Ve Güvenirliğinin İncelenmesi. Yüksek Lisans Tezi, Ege Üniversitesi.
- [Result] BENLİ M, YİĞİT KAYHAN N (2005). Ülkemizde Yaygın Kullanımı Olan Kekik (Thymus Vulgaris) Bitkisinin Antimikrobiyal Aktivitesi. Orlab On-Line Mikrobiyoloji Dergisi , 3(8) 1-8.
- [Result] Bardy J, Molassiotis A, Ryder WD, Mais K, Sykes A, Yap B, Lee L, Kaczmarski E, Slevin N. A double-blind, placebo-controlled, randomised trial of active manuka honey and standard oral care for radiation-induced oral mucositis. Br J Oral Maxillofac Surg. 2012 Apr;50(3):221-6. doi: 10.1016/j.bjoms.2011.03.005. Epub 2011 Jun 1. PMID 21636188
- [Result] Bardy J, Slevin NJ, Mais KL, Molassiotis A. A systematic review of honey uses and its potential value within oncology care. J Clin Nurs. 2008 Oct;17(19):2604-23. doi: 10.1111/j.1365-2702.2008.02304.x. PMID 18808626
- [Result] ATASOY, BESTE MELEK (2002). Radyoterapi Gören Baş Boyun Tümörlü Hastalarda Oluşan Akut ve Konik Kserostominin Amifostin ile Azaltılabilirliğinin İncelenmesi. Uzmanlık Tezi, Marmara Üniversitesi.
- [Result] ARSLANTAŞ TAMARA (2009). Kserostomi Oluşturulan Rat Modelinde Gastrik Reflünün Östaki Tüp Fonksiyonları Üzerine Olan Olumsuz Etkilerine Karşı Tükürüğün Koruyucu Etkileri. Uzmanlık Tezi, Süleyman Demirel Üniversitesi.
- [Result] Anggraeni DT, Hayati AT, Nur'aeni A. The effect of oral care using honey as an additional topical agent on oral health status of intubated patients in the intensive care unit. Enferm Intensiva (Engl Ed). 2022 Oct-Dec;33(4):225-232. doi: 10.1016/j.enfie.2021.12.004. PMID 36494157
- [Result] Bahramnezhad F, Dehghan Nayeri N, Bassampour SS, Khajeh M, Asgari P. Honey and Radiation-Induced Stomatitis in Patients With Head and Neck Cancer. Iran Red Crescent Med J. 2015 Oct 22;17(10):e19256. doi: 10.5812/ircmj.19256. eCollection 2015 Oct. PMID 26568850

DOCUMENTS (3):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT07358494/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT07358494/SAP_001.pdf
  • Informed Consent Form (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT07358494/ICF_002.pdf